CLINICAL TRIAL: NCT00847574
Title: Development, Implementation, & Testing and Education Program to Teach Weight Loss Using the 2005 Dietary Guidelines to Pre-Menopausal Women
Brief Title: The WORLD (Weight Optimization: Revamping Lifestyles Using the Dietary Guidelines) Study - Developing, Implementing, and Testing an Education Program
Acronym: WORLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WORLD Study; USDA CSREES #2005-55215-04811
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Cardiovascular Disease
Keywords: Weight loss; Weight maintenance; Weight management; Cardiovascular disease risk; Dietary Guidelines; Diet and exercise; Prevention
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate-fat (Experimental): 35% of calories from fat
  Interventions: Behavioral: Moderate-fat
- Lower-fat (Experimental): 20% of calories from fat
  Interventions: Behavioral: Lower-fat

INTERVENTIONS:
Behavioral: Moderate-fat — 35% of calories from fat
  Arms: Moderate-fat
Behavioral: Lower-fat — 20% of calories from fat
  Arms: Lower-fat

SUMMARY:
The WORLD study is a single-center, year-long randomized controlled trial in free-living women. Participants were randomly assigned to follow either a lower-fat (LF) diet or a moderate-fat (MF) diet for weight management in a parallel-arm design. The two phases of the study were a weight-loss phase (phase 1) and a weight-maintenance phase (phase 2) (Figure 1). During phase 1, months 1 through 4, participants consumed a hypo-caloric diet consistent with the 2005 Dietary Guidelines in the free-living environment. During phase 2, months 5 through 12, participants shifted into weight maintenance. It was hypothesized that a weight-loss intervention at the extremes of dietary fat recommendations of the 2005 Dietary Guidelines would be equally effective for weight loss while achieving comparable nutrient adequacy. Also, Overall, the lower-fat and moderate-fat diets would both be nutritionally adequate, based on the Healthy Eating Index.

ELIGIBILITY:
Inclusion Criteria:

* 21-50 years
* BMI: 25-39.9 kg/m2
* LDL-C: 100-189.9 mg/dL

Exclusion Criteria:

* Triglycerides > 350 mg/dL
* History of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease, and thyroid disease
* High alcohol consumption (<14 drinks/week)
* Use of medication or supplements for lowering blood lipid levels (i.e., statin, fibrates, psyllium, fish oil capsules, soy lecithin, phytoestrogens)
* Lactating, pregnant, or wanting to become pregnant during the study
* Weight loss or gain ≥ 10% body weight in the previous 6 months
* Eating Attitudes Test-26 score > 20
* Beck Depression Inventory-II score ≥ 29
* Gormally Cognitive Factors Related to Binge Eating Scale score > 30
* Physical Activity Readiness Questionnaire score > 2

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline, month 4, month 8, month 12

SECONDARY OUTCOMES:
Lipid Profile | Baseline, month 4, month 8, month 12
Glucose | Baseline, month 4, month 8, month 12
Insulin | Baseline, month 4, month 8, month 12
C-reactive protein | Baseline, month 4, month 8, month 12
Dietary intake | Baseline, month 4, month 12
Body composition | Baseline, month 4, month 12
Fitness via VO2max | Baseline, month 4, month 12
Cognitive-behavioral measures | Baseline, month 4, month 8, month 12

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, RD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.health.gov/DietaryGuidelines/